CLINICAL TRIAL: NCT05949255
Title: Probiotics and Insulin Resistance in Obese Asthmatics
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Lung Association (Other)
Responsible Party: Principal Investigator, Jessy S. Deshane, Associate Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-300011423; ALA 1143197 (Other Grant/Funding Number: American Lung Association Airways Clinical Research Network)
Record Dates: First submitted 2023-06-29; First posted 2023-07-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Asthma; Obesity; Insulin Resistance
MeSH Terms: conditions — Asthma; Obesity; Insulin Resistance | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Subjects will receive a probiotic supplement to take by mouth daily.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Subjects will receive a placebo to take by mouth daily.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — 10 subject will receive a probiotic daily for 12 weeks.
  Arms: Probiotic
Dietary Supplement: Placebo — 10 subjects will receive a placebo daily for 12 weeks.
  Arms: Placebo

SUMMARY:
In this pilot study investigators will test the hypothesis that administration of oral probiotics modulates microbiome/metabolome, lowers leptin and insulin resistance and improves clinical parameters of asthma in obese insulin resistant asthmatics. Preliminary studies with oral probiotic administration in obese asthmatics showed increased abundance of probiotics-derived Bifidobacterium species and Bifidobacterium-derived metabolite in the airways of asthmatics. Additionally, neutrophils and IL-17 producing Th17 cells were significantly reduced following probiotics administration. Based on these preliminary studies, the investigators propose to test the following aims:

Specific Aim 1: Determine if probiotic administration modulates airway microbiome/metabolome in obese insulin resistant asthmatics Specific Aim 2: Determine if modulation of leptin levels and insulin sensitivity by probiotics administration correlates with airway metabolome alterations and weight loss in obese insulin resistant asthmatics Specific Aim 3: Determine if microbiome/metabolome changes in probiotics group correlates with changes in asthma biomarkers and improved clinical outcomes compared to placebo in obese insulin resistant asthmatics.

DETAILED DESCRIPTION:
Participants for this study will be recruited through the UAB Asthma Clinic under an IRB approved protocol. The Asthma Clinic at UAB has over 350 unique patients. The composition of the clinic is 73% female, 58% non-hispanic white and 34% black/African American, and 63% have a BMI over 30. Asthma is defined by a constellation of symptoms including episodic dyspnea, cough, wheeze, and chest tightness with evidence of airway hyperresponsiveness. The subjects recruited to this study will be seen in the Asthma Clinic at UAB. All participants will have a clinical history of symptoms consistent with a diagnosis of asthma, and testing supporting the presence of airway hyperresponsiveness as denoted by either a positive bronchodilator response, a positive methacholine challenge test, or a high degree of clinical suspicion for asthma but unable to perform either of those tests. This study will recruit obese asthmatics with an Insulin Resistance score >5. Classification of obesity, waist circumference and waist-to-hip ratio (WHR) will be determined according to the WHO definitions. Body mass index (BMI kg/m2) of >30 will be considered obese. The Homeostatic model assessment (HOMA)-IR values >5 will be classified as those with severe IR. Additional patient information including age, sex, demographics and BMI will be collected at baseline and at 12 weeks. The HOMA-IR estimates steady-state β- cell function and insulin sensitivity and will be calculated by multiplying the fasting plasma glucose (mg/dl) value by serum insulin value (mIU/ml) value divided by 405. Potential participants will be prescreened for inclusion in this study. Patients in the Asthma Clinic who have previously agreed to participate in a local biorepository will have all of the prerequisite biometric data available, so only those individuals meeting inclusion criteria will be contacted for participation.

Participants (n=20 obese asthmatics) will be fasted for at least 12 hours prior to blood sampling at baseline. 20 obese asthmatic patients with BMI >30 and with IR >5 will be randomized and 10 patients will receive 1 capsule/day of 500 mg of probiotic supplement (Floragen Digestion, American Lifelines, Baraboo, WI ). This is a probiotic combination product ((Lactobacillus acidophilus, Bifidobacterium lactis, and Bifidobacterium longum (1.5 x 1010 CFUs/capsule)) and 10 patients in placebo group will receive 500 mg of starch per day for 12 weeks. For both study groups, both genders will be recruited equally with an anticipated distribution of approximately 40% African American and 60% Caucasian subjects. At baseline and at end of 12 weeks, respiratory function tests will be carried out and clinical endpoint measurements will be made. Additionally, nasal filters, nasal washes, rectal swabs, peripheral blood mononuclear cells and serum samples will be collected. 40 ml of peripheral blood samples will be collected at baseline and at 12 weeks after administration of probiotics or placebo control. These samples will be used for endpoint measurements in peripheral blood and serum. Microbiome analyses of nasal washes and rectal swabs will be carried out in collaboration with the UAB Microbiome core. For metabolomics studies, sampling of the upper airways of 60 participants with paired nasal filters and washes. The nasal filter method consists of introducing ~ 1/3 to 1/2 of a 15 × 25 mm filter paper made of synthetic absorptive matrix (Leukosorb, Pall Life Sciences) into one of the nostrils and placing it laterally against the anterior portion of the inferior nasal turbinate. The nasal filter will be left in the nostril for a minimum of 30 s and up to 2 min. Once removed, it will be placed into a sterile container. The nasal wash method consisted of using a bulb syringe to flush 3-5 mL of sterile, non-bacteriostatic, normal saline solution into the contralateral nostril. Both nasal filters and washes will be centrifuged and the supernatant transferred to a freezer and stored at - 80 °C until further processing.

ELIGIBILITY:
InclusionCriteria:

* Age > 18 years
* All patients will be obese asthmatics. Patients will have a body mass index >30 and insulin resistance>5.
* Asthmatics who have stable disease without changes to their asthma related medications for 3 months prior to enrollment

Exclusion Criteria:

* Asthma related hospitalization within 90 days of enrollment
* Asthma exacerbation requiring >3 days of oral corticosteroids within 28 days of enrollment
* Comorbid lung diseases other than asthma
* Pregnancy or planned pregnancy
* Inability to understand study procedures and/or provide informed consent
* Other significant medical conditions based on discretion of PI

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Determine if probiotic administration modulates airway microbiome/metabolome in obese insulin resistant asthmatics | 12 weeks
  (1a) For airway microbiome analyses, nasal wash samples will be used as surrogates. Nasal wash will be collected from subjects at baseline and 12 weeks. Rectal swab will be collected using Fecal swab kit (COPAN, Thermofisher) and samples prepared for microbiome analysis as above. Microbial genomic DNA from the samples will be isolated using the DNA isolation kit from Zymo Research.
  (1b) The samples obtained in Aim 1a will be used for metabolomics analyses, both gut and airway samples. Untargeted metabolomics utilizing Liquid Chromatography coupled with mass spectrometry will be performed at UAB Metabolomics Core and metabolites including SCFA, acetate, lactate, ethanol, succinate, formate and enterolactone will be analyzed and quantitated.
  For both above aims, changes over the 12 weeks will be compared between groups.
Determine if modulation of leptin levels and insulin sensitivity by probiotics administration correlates with airway metabolome alterations and weight loss in obese insulin resistant asthmatics | 12 weeks
  (2a) Classification of obesity, waist circumference and waist-to-hip ratio (WHR) will be determined according to the WHO definitions. At baseline and at 12 weeks post-probiotic administration, glucose, Leptin and lipid profile panels will be analyzed from plasma prepared from whole blood collected from fasting individuals.
  (2b) The recruited subjects will have a HOMA-IR >5. At baseline and at 12 weeks after probiotics/placebo administration, potential change in insulin sensitivity will be calculated as described in methods above. (2c) Determine if probiotic-mediated changes in leptin, weight gain and insulin sensitivity correlates with airway metabolome alterations compared to placebo controls. Unique airway metabolome signatures comparing probiotics and placebo control groups will be correlated with lowered leptin levels, increased weight loss and increased insulin sensitivity.
  For the above aims, changes over the 12 weeks will be compared between groups.
Determine if microbiome/metabolome changes in probiotics group correlates with changes in asthma biomarkers and improved clinical outcomes compared to placebo in obese insulin resistant asthmatics | 12 weeks
  (3a) At baseline and at 12 weeks post-probiotics or placebo administration, asthma biomarkers such as FeNO, IgE, peripheral neutrophils and eosinophils as well as proinflammatory plasma cytokines (IL-6, TNF-α, IL-1β) will be measured. Innate and adaptive immune cells will be enumerated by multiparameter flow cytometry in peripheral blood. These biomarkers will be correlated with changes in microbiome/metabolome identified above in Aim 1 between groups.
  (3b) At baseline and at 12 weeks post-probiotics or placebo administration, spirometry (FEV1 and FVC), exacerbations/steroid exposure, asthma control test (ACT) and asthma control questionnaire, Asthma Quality of Life Questionnaire (AQLQ) will be performed. Comparison in differences will be made between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jessy Deshane, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No